CLINICAL TRIAL: NCT00765505
Title: Muscle Lipid and Insulin Resistance in the Elderly
Acronym: MIRA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Erin E. Kershaw, M.D., Associate Professor, University of Pittsburgh
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0405764; 5R01AG021961 (NIH)
Record Dates: First submitted 2008-10-02; First posted 2008-10-03 (Estimated); Last update posted 2018-02-06 (Actual); Status verified 2018-02

CONDITIONS: Obesity
Keywords: Insulin Resistance; Obesity; Exercise Training; Physical Activity
MeSH Terms: conditions — Obesity; Insulin Resistance; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Exercise Group
  Interventions: Behavioral: Exercise Group
- Health Education Group (Experimental)
  Interventions: Behavioral: Health Education Group

INTERVENTIONS:
Behavioral: Exercise Group — Sixteen week intervention where subjects will be progressed to four days per week for 45 minutes per session, 180 minutes minimum per week, of moderate intensity supervised exercise.
  Arms: 1
Behavioral: Health Education Group — Sixteen week intervention. This group will not receive specific exercise education or prescription but will be asked to participate in biweekly health education sessions
  Arms: Health Education Group

SUMMARY:
This project will provide novel information concerning the ability of exercise to enhance the capacity for oxidative metabolism of fatty acids and improve insulin resistance in older adults who are at high risk for the development of type 2 diabetes. Ultimately this may help identify mechanisms and therapeutic targets implicated in skeletal muscle metabolic dysregulation. The proposed study is to conduct a randomized controlled exercise training intervention trial in older men and women. In addition, the response to exercise in these subjects will be compared to those of highly endurance-trained, age-matched athletes.

DETAILED DESCRIPTION:
Hypothesis and Specific Aims:

1. To determine whether aerobic exercise improves both skeletal muscle fat distribution and insulin sensitivity of older men and women. We will test two hypotheses.

   i. Physical exercise in older adults will decrease the amount of fat interspersed within muscle, specifically the fat between muscle groups (intermuscular adipose tissue) as well as decrease specific lipid metabolites within muscle cells, compared to controls.

   ii. Exercise-induced improvements in insulin sensitivity of older men and women will be related to the changes in muscle fat content independent of changes in total body fat or visceral abdominal adipose tissue.
2. To determine whether increased capacity for oxidative fatty acid metabolism within muscle results in improved insulin sensitivity in older adults. We will test two hypotheses.

   i. Exercise training will increase the capacity of muscle to oxidize fatty acids assessed both in vitro and in vivo.

   ii. Improved capacity for oxidative fatty acid metabolism will predict improvements in insulin sensitivity.

ELIGIBILITY:
Inclusion Criteria:

* 60 - 70 years of age
* No weight gain/loss of >10 lbs in 6 months
* Sedentary (No more than 1 continuous exercise/week) or Highly trained (>5 exercise sessions/week for a duration of one year or more)
* Non-Smoker
* BMI 18-38.0
* Resting blood pressure less than 150mmHg systolic/95 mmHg diastolic
* Normal glucose tolerance: Fasting glucose < 100 mg/dl or 2 hour glucose from OGTT < 140 mg/dl or impaired glucose tolerance (fasting glucose > 100 mg/dl < 126 mg/dl or 2 hour glucose from OGTT > 140 mg/dl but less than 200 mg/dl
* Note from PCP/Cardiologist for exercise clearance if positive stress test symptoms were observed from GXT

Exclusion Criteria:

* Clinically significant CVD including h/o MI
* Peripheral Vascular Disease
* Hepatic, renal, muscular/neuromuscular, or active hematologic/oncologic disease
* Clinically diminished pulse
* Presence of bruits in lower extremities
* Previous history of pulmonary emboli
* Peripheral Neuropathy
* Currently not engaged in a regular program and have a V)2 max pre-training value > 55 ml/kg-fat free mass-min., indicative of moderate fitness OR currently engaged in regular program and having a V)2 max value < 55 ml/kg-fat free mass-min.
* Anemia (Hematocrit < 34%)
* Any contraindications to moderate exercise
* Inability and/or willingness to comply with the protocol as written
* Active alcohol or substance abuse (Past 5 years)
* Total cholesterol > 300 mg/dL
* Triglyceride > 350 mg/dL
* ALT > 80, AST > 80, Alk Phos > 240
* Proteinuria (defined as > 1+ on routine dipstick) hypothyroidism (sTSH>8)
* Therapeutic Doses of Nicotinic Acid
* Type 2 Diabetes: Fasting Glucose > 126 mg/dl or 2 hour glucose > 200 mg/dl
* Oral Glucocorticoids
* Females currently on hormone replacement therapy (HRT) less than 6 months
* Claustrophobia
* Previous difficulty with lidocaine or other local anesthetic
* Stress test symptoms:

  * Positive ECG (>2mm ST segment depression) without PCP cardiologist permission to participate
  * Signs or symptoms of cardiovascular decomposition (hypotensive response to exercise
  * Onset of angina or angina like symptoms, shortness of breath, change in heart rhythm, signs of poor perfusion (light-headedness), tightness
  * Hypotension

Ages: 60 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 92 (Actual)
Dates: Start 2004-07; Primary Completion 2017-12-31 (Actual); Study Completion 2017-12-31 (Actual)

PRIMARY OUTCOMES:
Insulin sensitivity and muscle fat content will be measured at the beginning and the end of the intervention to determine the effects of exercise on these measures. | 16 weeks

SECONDARY OUTCOMES:
Examine if exercise-induced improvements in insulin sensitivity are similar in normal weight and in obese older subjects. | 16 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Bret H. Goodpaster, PhD, Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh, Pittsburgh, Pennsylvania, United States